CLINICAL TRIAL: NCT01905839
Title: A Longitudinal Study Assessing the Pathophysiology of Movement Disorders Utilizing the QMAT at Home Testing Device
Brief Title: A Study of Movement Disorders Using the QMAT At-Home Testing Device
Status: Terminated | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130167; 13-N-0167
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2015-04-15

CONDITIONS: Movement Disorders; Parkinson's Disease
Keywords: Rigidity; Assessment; Parkinson's Disease; Physiological Measures
MeSH Terms: conditions — Movement Disorders; Parkinson Disease; Muscle Rigidity

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Parkinson s disease (PD) affects half a million Americans, causing slow movements, tremors, stiffness, and trouble walking. Currently, these symptoms are measured by physical exam, but this is unreliable and requires an office visit. Researchers want to study a different way to measure PD symptoms, using a home-testing machine called a QMAT device. It can test how quickly someone moves doing different tasks. Researchers will study how this testing compares to physical exam testing and whether the device can detect changes in PD symptoms over time.

Objectives:

- To see if a home testing device can be used to evaluate Parkinson s disease symptoms.

Eligibility:

- Adults at least 18 years old with PD.

Design:

* Participants will have about 22 clinic visits over 5 years. Each visit will take up to 3 hours. Visits will be scheduled along with visits for another study.
* At visit 1, participants will learn to use the QMAT device and how to send testing information to the clinic by computer. The device has a computer screen, some buttons, and some pegs. Participants will get a device to take home and any accessories.
* Participants will learn 2 QMAT tests. For one, they will press keys as fast as possible. For the other, they will move pegs into holes. The tests will take a total of about 20 minutes.
* Participants will take both tests at home, 2 times on the same day each week, once before their medication, once after.
* A study coordinator will monitor the participant s computer data and discuss the at-home testing at the clinic visits.

DETAILED DESCRIPTION:
Objectives

The purpose of this protocol is to improve the understanding of the pathophysiology of movement disorders and to assess movement in Parkinson s disease by performing small behavioral exercises and objectively measuring movements utilizing the QMAT at home testing device. These devices will be provided by the Kinetics Foundation. We have developed a series of motor tasks that can be performed with the QMAT, a home-based computer module, so that data on patient s movement can be collected frequently and prospectively without obligating the patient to come to a medical center. The study is designed to be observational in nature.

The QMAT device is being implemented to respond to the interest in objectified tests to monitor, analyze, and further understand the physiological aspects of Parkinson s disease. We will conduct:

* Training to patients to perform tasks on the QMAT device and transmit data at home.
* Training to investigators who do not have prior experience using the system
* Testing using the QMAT device that may increase knowledge of a disease process, responsiveness of treatment or be helpful in patient progress evaluations by analyzing data collected from the at home tests.

This protocol includes only non-invasive techniques with minimal risk to the participants. The technique has been piloted as part of the 10-N-0009 protocol, Physiological Investigations in Movement Disorders.

Study Population

We intend to study patients with diagnosis of Parkinson Disease.

We will enroll up to 60 participants in order to obtain 48 patients who complete the study.

Design

We will assign and train study participants to use the QMAT device at home. This is a portable device with a simple keyboard and pegboard interface, storing data from patient performance at home. There are 2 tasks that are performed using the device. The pegboard task involves transferring pegs from holes on one side of the device to the opposite side of the device. The finger tapping test and the digitography tasks involve having the subject press keys on the keyboard. At enrollment into this study, a time schedule will be discussed with the participant regarding the schedule that these at home tests require to be conducted. We will provide the device, all the components, and a data storage thumb-drive to each participant.

Outcome measures

i. Bradykinesia (fine motor movements):

The component of the apparatus that will test fine motor control will involve finger pads that will be tapped in alternating fashion by the patient for 30 seconds.

The primary outcome variable will be mean keystroke velocity (completed alternating cycles/testing period, expressed as cm/sec. Secondary outcomes will be mean frequency expressed as Hz, mean strike duration, expressed as m/sec and temporal variation of the duration of finger strike and frequency (issues of fatigue) expressed as the coefficient of variation (SD/mean). Variation in velocity will be expressed as the SD.

ii. Complex movements: (Pegboard or plugging device):

The At-Home device also contains plugging tasks. Primary outcome: mean movement velocity expressed as seconds per plugging cycle. This measure can be analyzed statistically for all movements to correct for outlier responses and errors. A secondary outcome will also be defatigation (i.e., the linear change of speed during a testing session, expressed as percent of the cycle-time. The variance of speed will be provided by the standard deviation. A regression analysis will allow estimates of the part of the variance that is declared by linear change over the complete task.

ELIGIBILITY:
* INCLUSION CRITERIA
* Patients will have a diagnosis of Parkinson Disease
* Age 18 or older
* Able to give informed consent
* Ability to comply by the schedule and routine of taking the at home tests with the QMAT system responsibly
* ability to perform the QMAT testing
* current or planned enrollment in 12-N-0137: A Phase 1 Open-label Dose Escalation Safety Study of Convection-Enhanced Delivery (CED) of Adeno-Associated Virus Encoding Glial Cell Line-Derived Neurotrophic Factor (AAV2-GDNF) in Subjects with Advanced Parkinson s Disease

EXCLUSION CRITERIA

* Have more than 7 alcoholic drinks a week in the case of a woman or 14 alcoholic drinks a week in the case of a man.
* Have had a brain tumor, a stroke, head trauma, epilepsy, or a history of seizures.
* Have major depression or any major mental disorders (axis I disorders).
* Have other neurologic disorder than a movement disorder
* Have had a head injury where there was a loss of consciousness for more than a few seconds.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-06-18; Primary Completion 2015-04-15 (Actual); Study Completion 2015-04-15 (Actual)

PRIMARY OUTCOMES:
Mean speed of keystrokes on a repetitive finger movement | 5 years follow up
Mean speed of movement on a peg movement task | 5 years follow up

CONTACTS AND LOCATIONS:
Overall Officials: Codrin I Lungu, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Adler CH, Hentz JG, Joyce JN, Beach T, Caviness JN. Motor impairment in normal aging, clinically possible Parkinson's disease, and clinically probable Parkinson's disease: longitudinal evaluation of a cohort of prospective brain donors. Parkinsonism Relat Disord. 2002 Dec;9(2):103-10. doi: 10.1016/s1353-8020(02)00012-3. PMID 12473400
- [Background] Bronte-Stewart HM, Ding L, Alexander C, Zhou Y, Moore GP. Quantitative digitography (QDG): a sensitive measure of digital motor control in idiopathic Parkinson's disease. Mov Disord. 2000 Jan;15(1):36-47. doi: 10.1002/1531-8257(200001)15:13.0.co;2-m. PMID 10634240
- [Background] Muller T, Benz S. Quantification of the dopaminergic response in Parkinson's disease. Parkinsonism Relat Disord. 2002 Jan;8(3):181-6. doi: 10.1016/s1353-8020(01)00010-4. PMID 12039429